CLINICAL TRIAL: NCT00954551
Title: Utility of Serum Procalcitonin Levels to Distinguish Systemic Inflammatory Response From Systemic Infection in Febrile Subarachnoid Hemorrhage Patients
Brief Title: Serum Procalcitonin
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Emir Festic, M.D., Mayo Clinic
Other Study IDs: 09-000909
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Subarachnoid Hemorrhage (SAH)
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All adult patients with SAH in ICU: All adult patients admitted for an expected ICU stay of more than 24 hrs over a 6-month period (tentative) between xx and xx 2009 with a diagnosis of SAH will be prospectively evaluated.

SUMMARY:
Systemic inflammatory response syndrome (SIRS) is characterized by changes in body temperature, heart rate, respiratory rate, or peripheral blood white cell count, and is often a heralding manifestation of blood infection (ie., sepsis or bloodstream infection). SIRS however can occur as a result of a stroke without sepsis. When SIRS occurs after stroke, patients are subjected to blood cultures and tests to exclude sepsis, and are often empirically treated with antibiotics potentially leading to a serious gastrointestinal infection called C. difficile enterocolitis, and bacterial antibiotic resistance. Development of a blood test that could provide sufficient sensitivity to exclude blood infection in stroke would therefore prevent numerous tests, cultures, antibiotics, and costs. In recent years, there has been increasing evidence that procalcitonin (PCT) may serve as diagnostic marker to distinguish between infectious and non-infectious SIRS. The investigators hypothesize that PCT can differentiate SIRS after stroke into patients with infection and those without infection. Such screening tests would provide crucial information to clinicians that could improve patient care by reducing the number of tests and antibiotics used, as well as antibiotic-related infections, bacterial resistance and hospital costs.

Hypothesis: The investigators hypothesize that PCT can be used to define normal (SIRS without infection) and abnormal values SIRS with infection (i.e., blood, lung, urinary, spinal fluid) in a population of patients with aneurysmal subarachnoid hemorrhage (SAH).

Specific Aim 1.) To establish normal values of PCT in patients with aneurysmal subarachnoid hemorrhage and SIRS.

Specific Aim 2.) Derive the sensitivity and positive predictive value of abnormal PCT values in patients with aneurysmal SAH, SIRS with true systemic infection.

DETAILED DESCRIPTION:
Hypothesis: We hypothesize that PCT can be used to define normal (SIRS without infection) and abnormal values SIRS with infection (i.e., blood, lung, urinary, spinal fluid) in a population of patients with aneurysmal subarachnoid hemorrhage (SAH).

Specific Aim 1.) To establish normal values of PCT in patients with aneurysmal subarachnoid hemorrhage and SIRS.

Specific Aim 2.) Derive the sensitivity and positive predictive value of abnormal PCT values in patients with aneurysmal SAH, SIRS with true systemic infection.

Stroke is the third leading cause of death in the United States (AHA), A ruptured brain aneurysm leads to subarachnoid hemorrhage (SAH) which is a common but deadly stroke subtype (8% of all strokes). SAH one-month mortality is at least 30-40% from a combination of complications, being either cerebral (seizures, re-bleeding, hydrocephalus, herniation, coma, brain death) or extra-cerebral (pulmonary edema, myocardial stunning/infarction, hyponatremia, and SIRS). SIRS after subarachnoid hemorrhage is common, and is associated with the increased mortality of SAH (Yoshimoto Y). The pathogenesis remains of SIRS after SAH remains poorly understood, but theorized to be a results of catecholamines (e.g., adrenaline) and interleukins leading to increased heart and respiratory rate, increased peripheral white blood cell count and fever (Wartenberg K). Therefore SIRS after SAH mimics true systemic infection (e.g., sepsis) even when no true infection exists. Lack of treatment of true infection in SAH patients for presumptive non-infective SIRS can lead to missed sepsis and death.

* A prospective, observational study is proposed
* PCT levels will be obtained with daily intensive care unit laboratory values on the initial day (day #1), day 3, 5, 7, 9, 11, and 13.
* Patients with presumed infection will have the following comprehensive assessment per ICU standard of care when a SAH patient has a fever (i.e., temperature 38.5 oral or greater or 38.0 core temperature or greater): two sets of peripheral blood cultures, one cerebrospinal fluid (CSF) culture,

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted for an expected ICU stay of more than 24 hrs over a 6-month period

Exclusion Criteria:

* Patients with known hyper-bilirubinemia (>0.4 mg/ml) or hypertriglyceridemia (>10 g/l) will be excluded since this can interfere with measurements of PCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted for an expected ICU stay of more than 24 hrs over a 6-month period (tentative) between xx and xx 2009 with a diagnosis of SAH will be prospectively evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
All adult patients admitted for an expected ICU stay of more than 24 hrs over a 6-month period (tentative). | 6 months

SECONDARY OUTCOMES:
SIRS criteria require 2 or more of the following variables (SCCM reference): 1.) alternations in body temperature 2.) alteration in peripheral white blood cell count 3.) tachycardia 4.) respiratory rate of more than 20 breaths per minute | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Emir Festic, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States